CLINICAL TRIAL: NCT06306404
Title: The Role of Online Sleep Intervention and Hormone Therapy on Sleep, Climacteric Symptoms and Mood in the Perimenopause
Brief Title: Sleeping Through Menopause
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Birit Broekman, Prof. dr. MD, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-512071-12-00
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Menopause; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Estrogens; Progestins; Hormone Replacement Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- MHT (Experimental): Participants will receive the standard care menopausal hormone therapy.
  Interventions: Drug: Estrogens and Progestogens
- Sleep modules (Experimental): Participants will receive the sleep modules, which includes cognitive behavioral therapy for insomnia, and circadian rhythm therapy.
- MHT and Sleep modules (Experimental): Participants will receive both the sleep modules, which includes cognitive behavioral therapy for insomnia, and circadian rhythm therapy, and the standard care menopausal hormone therapy.
  Interventions: Drug: Estrogens and Progestogens; Behavioral: Cognitive behavioral therapy for insomnia (CBTi), and circadian rhythm therapy
- No intervention (No Intervention): The control group.

INTERVENTIONS:
Drug: Estrogens and Progestogens — Menopausal Hormone Therapy, formerly known as Hormone Replacement Therapy (HRT), is a medical treatment that involves the use of hormones to relieve the symptoms of menopause and to reduce the risk of certain long-term health conditions associated with menopause. Menopause is a natural biological process that occurs when a women's ovaries stop producing effects, and her estrogen and progesteron hormone levels subsequently decrease. MHT typically involves administration of a combination of sec steroids.
  In this study MHT consists of estradiol transdermal patches (50 mcg (Systen), which provide a stable release of estradiol and lead to more stable blood levels. This is combined with 200 mg progesterone (Utrogestan tablets for 2 weeks) adjusted to the menstrual cycle to prevent endometrium carcinoma according to the international MHT guidelines.
  Other Names: Hormone replacement therapy
  Arms: MHT; MHT and Sleep modules
Behavioral: Cognitive behavioral therapy for insomnia (CBTi), and circadian rhythm therapy — CBTi is a guided, internet-based cognitive behavioral therapy program for insomnia, containing information and exercises on sleep. It consists of five online sessions:
  1. Psycho-education on sleep, disordered sleep and sleep hygiene (i.e. general guidelines about health and environmental factors influencing sleep),
  2. Sleep restriction (i.e. restrict time in bed to the average sleep time) and stimulus control training (i.e. reinforce association of bed with sleeping),
  3. Rumination and relaxation techniques,
  4. Cognitive restructuring (i.e. changing misconceptions about sleep),
  5. Relapse prevention.
  Arms: MHT and Sleep modules

SUMMARY:
Sleepless nights during the menopausal period: what treatment works? About half of the women have trouble sleeping during the years around the menopause, the perimenopause. This is a period characterised by fluctuating sex hormones. Insomnia during the perimenopause can make women more likely to develop more severe climacteric symptoms and other mental health problems. It is therefore important to find the right treatment to treat insomnia. Currently, we do not know what the best treatment is for managing insomnia during the perimenopause. The Sleeping Through Menopause study is the first to evaluate, side by side, two interventions: menopausal hormone therapy (MHT) and combined cognitive behavioural and circadian therapy for insomnia (CBCTi). The study aims to evaluate how well these treatments alleviate insomnia and climacteric symptoms including hot flashes, and by doing so alleviate or prevent other mental health issues. It will also explore how personal factors might affect treatment success.

In the study, 222 women with both insomnia and climacteric symptoms will be randomly assigned to one of four groups: MHT, CBCTi, a combination of both MHT and CBCTi, or a group with no treatment. The main goal is to evaluate how each treatment alleviates insomnia after 8 and 15 weeks. Secondary outcomes are sleep quality, climacteric symptoms including hot flashes, mental health, and daily functioning.

This study will help us understand the best ways to treat sleep problems during menopause and whether better sleep can improve other mental health and menopausal symptoms as well.

DETAILED DESCRIPTION:
The perimenopause is known as a vulnerable period for some women, with noticeable somatic and psychological issues. Aside from climacteric symptoms, insomnia and depression are common. About half of women during the peri-menopausal period experience sleep problems like problems falling asleep, awakening during the night and being unable to return to sleep. This is often attributed to vasomotor symptoms, but this is not the only reason of poor sleep. Also, the peri-menopausal period is a critical time for the occurrence of new onset and recurrent depressions. It has been suggested that fluctuations in estradiol may increase the risk for depression by altering neuronal functions in the brain. But there are also indications that the risk for depression increases by indirect effects, such as the increase in insomnia. Poor sleep has increasingly been recognized as the key modifiable factor affecting mental issues like depression. While antidepressants and psychotherapies continue to be the treatments of choice for depression, and Cognitive Behavioral Therapy for sleep (CBTi) for insomnia, preclinical and clinical data support the benefits of estrogen-based therapies to improve mood, sleep and other menopause-related symptoms. Transdermal estradiol patches, which provide a stable release of estradiol and lead to more stable blood levels, have been suggested to have a positive effect on sleep and depressive symptoms in randomized controlled trials. However, it is currently unclear if the relation between improvement in mood and estradiol patches is mediated by improvement in sleep problems, and if the effect of estradiol patches on sleep problems is more effective during peri-menopause than the current evidence-based sleep interventions of CBTi, preferably in combination with Circadian Rhythm Support (CRS). The aim of the study is to pinpoint the determinants of complaints about sleep and mood and how they respond to Menopausal Hormone Treatment (MHT) with and without the addition of a guided eHealth sleep intervention that combines CBTi + CRS.

Measurements will be conducted at baseline (T0), 2 months (T1) and 4 months (T3), with questionnaires, sleep measurements (EEG sleepband and actigraph) and skin conductance (to measure hot flushes). Participants will be recruited via www.slaapregister.nl and via OLVG outpatient clinic population of peri-menopausal women seeking help for climacteric complaints (like hot flushes, feeling bloated, increase in weight), including sleep problems. The participants are adults between 40-55 years old, with an Insomnia Severity Index score ≥10 and Climacteric Green Scale score ≥ 13.They have the self-considered capability to complete online questionnaires and diaries in Dutch.

The intervention will be MHT (estradiol transdermal patches 50 mcg (Systen), in combination with 200 mg progesterone (Utrogestan tablets for 2 weeks, adjusted to the menstrual cycle to prevent endometrium carcinoma according to the international MHT guidelines), with and without the addition of a guided eHealth sleep intervention that combines CBTi + CRS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40-55 years old
* Insomnia severity index score =>10
* Green Climacteric Score =>13
* Self-considered capability of completing online questionnaires and diaries in Dutch/English
* Presence of a menstruation (whether regular or not) and the last menstruation must be less than 12 months ago

Exclusion Criteria:

* CBTi treatment in past year
* Bipolar disorder or psychotic disorder
* Contra-indication for Menopausal Hormone Therapy
* Alcohol or drugs dependency (scores of ≥ 20 on the AUDIT and ≥25 on the DUDIT)
* Women using thyroid medication, lamotrigine, aromatase, tamoxifen, because of interaction effects with MHT
* Use of drugs known to interfere with cytochrome P450 enzyme (CYP) 3A4
* Known hypersensitivity to the excipients in the estradiol patch: acrylate copolymer, polyethylene terephthalate, alfa-tocopherol, soy allergy (component of progesterone capsule).
* All women on hormonal contraceptives will be excluded.
* All women already on MHT will be excluded.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable is the difference between the groups in the within-subject change in insomnia severity at T1 (2 months) and T2 (4 months) relative to T0 (baseline). | month 2 vs. month 4
  The Insomnia Severity Index (ISI) is composed of seven items that evaluate the severity of sleep disturbance during the past 2 weeks. Each item is rated on a five-point Likert scale and the total score indicates the severity of insomnia. The higher the more severe.

CONTACTS AND LOCATIONS:
Overall Officials: Birit Broekman, Prof., Principal Investigator — OLVG and Amsterdam UMC, VU; Eus van Someren, Prof., Principal Investigator — Netherlands Institute for Neuroscience

IPD SHARING:
Plan to Share IPD: Yes